CLINICAL TRIAL: NCT06717633
Title: Comparison of Short-term Effects of Extracorporeal Shock Wave Therapy, Low-level Laser Therapy and Pulsed Electromagnetic Field Therapy in Knee Osteoarthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, Medical Doctor, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: modalities
Record Dates: First submitted 2024-11-30; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Extracorporeal Shockwave Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control (No Intervention): Control group only receives a daily exercise program, including knee joint range of motion, stretching, and strengthening exercises.
- ESWT (Experimental): The ESWT will be administered using an ESWT device (Modus ESWT Compact Model-Portable) once weekly over three consecutive weeks, resulting in a total of three sessions. A radial shockwave mode was chosen for the therapy. During each session, participants will receive 3000 pulses at an 12-Hz frequency and pneumatic pressure of 2.5 bars
  Interventions: Device: extracorporeal shock wave therapy
- LLLT (Experimental): The MLS (Multiwave Locked System) laser is a specific type of low-level laser therapy (LLLT) that combines two different wavelengths of light-typically 808 nm (near-infrared) and 905 nm (mid-infrared)-to produce therapeutic effects. These wavelengths are delivered simultaneously in a synchronized manner, which is intended to enhance the overall effectiveness of the treatment. LLLT will be conducted with the laser device (MLS Laser M6 Robotic Multiwave Lock System, Asalaser, Italy) with the use of protective goggles, and the treatment parameters were set as follows: 100% power, 3 Joules per treatment spot with 904 nm wavelength, and a treatment area of 20 cm². The LLLT will be applied to five points on the anterior part of the joint space, with each point treated for 3 minutes, totaling 15 minutes. A total of 8 sessions were applied for 4 weeks, 2 days a week.
  Interventions: Device: low-level laser therapy
- PEMF (Experimental): For PEMF, the applicator of the device (Easy QS Magnetotherapy Portable Magnetotherapy Medical Device, Asalaser, Italy) will be positioned to target the medial and lateral aspects of the knee. The treatment parameters were defined as follows: rectangular field shape, 30 Hz frequency, 10 mT intensity, and a duration of 20 minutes. A total of 8 sessions were applied for 4 weeks, 2 days a week.
  Interventions: Device: pulsed electromagnetic field therapy

INTERVENTIONS:
Device: extracorporeal shock wave therapy — The ESWT will be administered using an ESWT device (Modus ESWT Compact Model-Portable) once weekly over three consecutive weeks, resulting in a total of three sessions. A radial shockwave mode was chosen for the therapy. During each session, participants will receive 3000 pulses at an 12-Hz frequency and pneumatic pressure of 2.5 bars
  Arms: ESWT
Device: low-level laser therapy — The MLS (Multiwave Locked System) laser is a specific type of low-level laser therapy (LLLT) that combines two different wavelengths of light-typically 808 nm (near-infrared) and 905 nm (mid-infrared)-to produce therapeutic effects. These wavelengths are delivered simultaneously in a synchronized manner, which is intended to enhance the overall effectiveness of the treatment. LLLT will be conducted with the laser device (MLS Laser M6 Robotic Multiwave Lock System, Asalaser, Italy) with the use of protective goggles, and the treatment parameters were set as follows: 100% power, 3 Joules per treatment spot with 904 nm wavelength, and a treatment area of 20 cm². The LLLT will be applied to five points on the anterior part of the joint space, with each point treated for 3 minutes, totaling 15 minutes. A total of 8 sessions were applied for 4 weeks, 2 days a week.
  Arms: LLLT
Device: pulsed electromagnetic field therapy — For PEMF, the applicator of the device (Easy QS Magnetotherapy Portable Magnetotherapy Medical Device, Asalaser, Italy) will be positioned to target the medial and lateral aspects of the knee. The treatment parameters were defined as follows: rectangular field shape, 30 Hz frequency, 10 mT intensity, and a duration of 20 minutes. A total of 8 sessions were applied for 4 weeks, 2 days a week.
  Arms: PEMF

SUMMARY:
120 patients with Kellgren-Lawrence grade 2-3 knee osteoarthritis will be randomized into four groups: Control group, Extracorporeal shock wave therapy (ESWT) (once a week for 3 sessions), Low-level laser therapy (LLLT) (twice a week for 8 sessions), and Pulsed electromagnetic field therapy (PEMF) (twice a week for 8 sessions), with 30 patients in each group. All participants will be instructed in a daily exercise program, including knee joint range of motion, stretching, and strengthening exercises (3×10 repetitions). Outcome measures, including the Visual Analogue Scale (VAS), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), Short Form-36 (SF-36), and Timed Up & Go (TUG) test, will be assessed at baseline after treatment and at 3rd month.

ELIGIBILITY:
Inclusion Criteria:

* experiencing knee pain persisting for more than 6 months, radiological assessment confirming grade 2 and grade 3 knee osteoarthritis based on the Kellgren-Lawrence system
* no history of physical therapy or regular use of non-steroidal anti-inflammatory drugs (NSAIDs) within the last 6 months,
* absence of any pathology other than osteoarthritis that could cause knee pain,
* no lumbar spine or hip pathology that could refer pain to the knee,
* free from any conditions that would prevent participation in exercise or physical therapy
* willing to regularly participate the treatment programs were included in the study.

Exclusion Criteria:

* presence of a condition that impairs ambulation,
* a documented history of spinal stenosis,
* evidence of a neurological disorder based on medical history or physical examination,
* the existence of an inflammatory or metabolic disorder that could lead to secondary osteoarthritis,
* administration of intra-articular knee injections within the past year,
* use of NSAIDs, paracetamol or topical agents within the preceding week,
* a prior history of surgical intervention involving the knee joint.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-27 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | baseline after treatment and at 3rd month
  Pain assessment in the study was conducted using the VAS, which ranges from 0 to 10. Patients were instructed to evaluate the pain they experienced. A score of "0" signified the absence of pain, whereas a score of "10" denoted the most intense pain they had ever encountered in their lifetime.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline after treatment and at 3rd month
  The WOMAC OA Index is a questionnaire completed by the patient to assess pain, stiffness, and physical function related to knee and hip osteoarthritis. It consists of 24 questions addressing pain, stiffness, and physical function. The index provides both a total score and separate subscores for each category. Higher scores indicate poorer outcomes in that category.
Short Form-36 (SF-36) | baseline after treatment and at 3rd month
  Among quality of life scales, the SF-36 is a generic scale that provides a broad assessment. It comprises 36 items that assess eight dimensions: physical functioning (PF), social functioning (SF), role limitations due to physical health (RLPH), role limitations due to emotional problems (RLEP), emotional well-being (EW), energy/fatigue (E), pain (P), general health (GH) and health change (HC).
Timed Up & Go Test (TUG) | baseline after treatment and at 3rd month
  This test is designed to assess dynamic balance and functional mobility. The test requires a chair, a stopwatch, and a 3-meter walking space. It begins with the individual seated in a chair. Upon receiving the instruction, the individual stands up, walks 3 meters at a regular speed, turns around, walks back to the starting point, and then sits down again. The time taken to complete the test is recorded in seconds for scoring purposes.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Goztepe Prof Dr Suleyman Yalcin City Hospital, Istanbul, None Selected, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No